CLINICAL TRIAL: NCT05948098
Title: The Effect of Facilitated Tucking Position and Gentle Human Touch Practices on the Perception of Pain During Heel Blood Collection in Premature Newborns
Brief Title: Facilitated Tucking Position, Gentle Human Touch Practices and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Tuba Koc Ozkan, Associate professor, Adiyaman University Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HRÜ/230818
Record Dates: First submitted 2023-06-30; First posted 2023-07-17 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Pain; Premature
MeSH Terms: conditions — Pain; Premature Birth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Facilitated Tucking Position (Experimental): Prior to the procedure, parents will be informed about facilitated tucking position practices.Heel blood will be drawn from newborns after facilitated tucking position practices are performed. The pain of newborns will be evaluated with the "Neonatal Pain Diagnostic Scale (NIPS)" before, during and after the procedure. Practice:
  For the facilitated tucking position, the lower and upper extremities of the newborn will be kept in lateral flexion and close to the midline. Meanwhile, the researcher's hand will be gently held on the baby's head and the other hand on the baby's hips, without restricting the baby's movements. The facilitated tucking position will be given one minute before the heel blood collection and will be maintained for one minute during and after the blood collection.
  Interventions: Behavioral: Facilitated Tucking Position
- Gentle Human Touch (Experimental): Before the procedure, parents will be informed about gentle human touch practice. After Gentle human touch practice, heel blood will be taken from newborns. The pain of newborns will be evaluated with the "Neonatal Pain Diagnostic Scale (NIPS)" before, during and after the procedure. Practice:
  For the Gentle human touch practice, the researcher will place one hand on the newborn's top (head) above the brow line and the other hand on the lower abdomen covering the baby's waist and hips. Gentle human touch practice will be started 10-15 minutes before the procedure and will continue throughout the process and until 15 minutes after the end of the process.
  Interventions: Behavioral: Gentle Human Touch
- Control Group (No Intervention): During the heel blood collection, no procedures other than routine procedures applied in the clinic will be applied. The pain of newborns will be evaluated with the "Neonatal Pain Diagnostic Scale (NIPS)" before, during and after the procedure.

INTERVENTIONS:
Behavioral: Facilitated Tucking Position — a sub-form of method of nesting the baby and the procedure of bringing the body to middle or even close position by holding the upper and lower extremities of the baby in flexion with hands
  Arms: Facilitated Tucking Position
Behavioral: Gentle Human Touch — It is a form of healing touch
  Arms: Gentle Human Touch

SUMMARY:
This prospective study is planned as a randomized controlled study to evaluate the effect of facilitated tucking position and gentle human touch practices on the pain experienced by newborns during heel blood collection. This study is planned to be carried out between 15 July and 15 December 2023 in the neonatal intensive care unit of a training and research hospital in the Southeastern Anatolia Region. The sample size was calculated based on the study of premature infants to determine the effect of facilitated tucking position on procedural pain. According to the results of the study, PIPP pain scores were determined as 11.88±3.05 in the intervention group (n=17) and 9.06±2.95 in the control group (n=17). The effect size of the study was determined as d= 0.939 at α=0.05 level and 95% confidence interval. It was decided to conduct the study with a total of 90 premature babies, 30 of whom were in the groups, in case of data loss during the study.

DETAILED DESCRIPTION:
Neonatal pain negatively affects prognosis, behavior, environmental adaptation, development of the brain and senses, and interaction. Effective management of neonatal pain supports health and recovery, shortens hospital stays, and reduces care costs and the prevalence of neurobehavioral problems. Therefore, proper management of pain in newborns is important for the healthy development of newborns. Many invasive procedures are applied to newborns hospitalized in neonatal intensive care units. Non-nutritive sucking, oral sucrose, kangaroo care, facilitated tucking position, and gentle human touch have proven to have positive effects on the pain experienced by newborns during interventional procedures. In this study, the effect of facilitated tucking position and gentle human touch practices applied during heel blood collection on the perception of pain in premature newborns will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborns (34-37 weeks of gestation), dependent on nasal CPAP, without congenital anomalies, not taking sedative or analgesic drugs, not receiving oral feeding, and whose parents approved to participate in the study will be included in the study.

Exclusion Criteria:

* Newborns with open wounds on their body, bleeding disorders, and those who underwent a painful procedure just before heel blood sampling will not be included in the study.

Ages: 34 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Neonatal Pain Diagnostic Scale (NIPS) | 1 minutes
  It was developed by Lawrence et al. in 1993 to evaluate interventional pain in newborns (Lawrence et al, 1993). Its Turkish adaptation was made by Akdovan and Yıldırım in 1999. NIPS is an assessment tool that focuses on six behavioral responses of newborns: facial expressions, crying, breathing, arm movements, leg movements, and arousal. A score between 0 and 7 is obtained from the scale, and as the score obtained from the scale increases, the pain of newborns also increases. In the Turkish adaptation study of the scale, the Cronbach's alpha value was calculated as 0.83 before the procedure, 0.83 during the procedure and 0.86 after the procedure.

SECONDARY OUTCOMES:
Pulse Oximeter Device | 1 minutes
  It was used for the measurement of oxygen saturation and heart rate before, during and after heel lancing in all three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Koç Özkan, Principal Investigator — Adiyaman University
Locations (1):
- Adıyaman University, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No